CLINICAL TRIAL: NCT02287506
Title: The StartRIGHT Pilot Study; Getting the Right Classification and Treatment From Diagnosis in Adults With Diabetes
Brief Title: StartRIGHT: A Pilot Research Study About Diabetes Diagnosis & Treatment
Acronym: StartRIGHT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot feasibility for full trial: NCT03737799
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRF166
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2015-02

CONDITIONS: Diabetes
Keywords: diagnosis, strategy
MeSH Terms: conditions — Diabetes Mellitus; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ODS from enrolment (Experimental): Optimised Diagnostic Strategy used from enrolment to study
  Interventions: Other: Optimised Diagnostic Strategy
- ODS at end of study (No Intervention): ODS fed back at the end of the participants involvement with the study

INTERVENTIONS:
Other: Optimised Diagnostic Strategy — (ODS) based on integrating Clinical information (a validated clinical probability model), Biomarkers (GAD, IA2 and ZnT8 autoantibodies) and Genetic testing for MODY
  Other Names: ODS
  Arms: ODS from enrolment

SUMMARY:
This study aims to achieve more accurate early classification of diabetes and identification of which patients will rapidly require insulin treatment. The investigators will recruit 1000 participants who have been diagnosed with diabetes in the last year and were aged between 18 and 50 years at the time of diagnosis. The investigators will recruit an additional cohort of 400 participants diagnosed after age 50 treated with insulin at recruitment. The investigators will record clinical features and biomarkers that may help us to determine diabetes type at diagnosis and follow participants for 3 years to assess the development of severe insulin deficiency (measured using C-peptide) and insulin requirement. The investigators will assess utility of clinical features and additional biomarkers in identifying patients with rapid progression to insulin requirement. Findings will be integrated into a freely available clinical prediction model.

DETAILED DESCRIPTION:
Diabetes is stratified into recognised subtypes with major implications for patients' treatment. The treatment of Type 1 diabetes (T1D), Type 2 diabetes (T2D) and Maturity-onset diabetes of the young (MODY) is markedly different and based on clear differences in underlying pathophysiology. The difficult part of this stratification is correctly diagnosing the subtype especially in young adults. The clear differentiation of T1D as slim and young, and T2D as obese and old, no longer holds with the rapid increase in obesity in the population: T1D patients may be obese and T2D patients may be diagnosed young. 90% of MODY patients are misdiagnosed with T1D or T2D as the diagnosis of MODY is rarely considered. This results in 7-15% of young adults with diabetes being wrongly classified and incorrectly treated. Initial clinical diagnosis is not systematic and once made is rarely changed. Misdiagnosis of T2D or MODY as T1D results in unnecessary initial insulin treatment leading to higher drug/monitoring costs, more side effects (weight gain, hypos), and patient inconvenience/dissatisfaction. Misdiagnosis of T1D as T2D, or MODY (initial treatment diet/tablets), results in poor glycaemic control, frequent contact for increased treatment, inappropriate insulin regimes and the risk of life threatening ketoacidosis.

The investigators have developed an optimized diagnostic strategy (ODS) based on integrating Clinical information (a validated clinical probability model), Biomarkers (GAD, Islet antigen-2 (IA2) and ZnT8 autoantibodies) and Genetic testing for MODY. This has the potential to determine the subtype of diabetes in young adults leading to improved treatment and care. Prior to undertaking a comprehensive RCT to test our ODS against standard care, the investigators must first undertake this pilot study to assess the feasibility of such a project.

Objectives: To assess the feasibility of recruitment and retention for a proposed large scale RCT, optimize recruitment and retention strategies, develop and assess the protocols and procedures, test delivery of the ODS, assess the impact of the ODS and obtain pilot data to inform sample size calculations for the proposed RCT Potential participants will be identified from routine clinical care, with clinicians informing patients of the project in general terms and seeking permission for their contact details to be passed to the research team. A range of referral strategies will be assessed and all potential participants who appear to meet the entry criteria will be invited to participate.

Referral strategies to be assessed will include: referral to research team by GP/ Practice Nurse/diabetes specialist nurse, regular GP practice database searches, via pathology lab following raised Hba1c Initial visit (I hour): Participants will meet with a member of the research team who will obtain consent and collect baseline blood samples, demographic and QoL data. Participants will be randomised to either the intervention or control arm using a computer generated randomisation schedule. For participants in the intervention arm the blood samples will be analysed at the Royal Devon &Exeter National Health Service Foundation Trust (RD&E NHS FT) Biochemistry Department for HbA1c, C-peptide and islet autoantibodies (GAD, IA2 and ZnT8) with DNA extracted and stored for genetic testing if appropriate. These blood results will then be immediately incorporated into the ODS for feedback to Clinicians and participants with recommendations that appropriate national guidelines for the ODS diagnosis (e.g. NICE guidelines for Type 1 or Type 2 diabetes) are followed. For participants in the control arm their current clinical features will be recorded and their blood samples will be stored for future analysis. At the end of their involvement in the study, both recorded clinical features and results from stored blood samples will then be and incorporated into the ODS for feedback to both clinicians and participant.

Follow up (6 monthly intervals over 3 years): Participants will then be followed up at 6 monthly intervals over a 3 year period (choice given of text, phone, or email) to maintain participant engagement and enable collection of details of current treatment, treatment changes and frequency of hypoglycaemia. Results from routinely collected HbA1cs will be obtained from clinical practice.

At 3 years, participants will be seen again by the research team for collection of a further blood sample, details of final treatment and quality of life measures. This will end their participation. At the end of the study individual results from the ODS for those in the control (standard care) arm will be generated and fed back to clinicians and participants.

All participants will be assigned a unique study ID. All data collected will be recorded and stored under this ID number. Data will be initially recorded onto a study specific data collection form (DCF). Data will then be recorded onto a study specific database. Hard/scanned copies will be stored in the study specific site file. Data will be screening for discrepancies and missing data prior to analysis.

Baseline data will include: personal identifiers, anthropometry, diabetes and medication history and blood biochemistry. Permission will be obtained to access medical notes should this be required for diabetes data relevant to taking part in the project.

All participant data will be held in a link-anonymised format, Participants' research and sample data will be identified by unique study ID numbers and all data will be held on password-protected computers. Only the CI or designated research team member will have access to personal identifiable data.

Data Storage and Archiving: All consent and paper data collection forms will be scanned onto discs and stored in locked filing cabinets within the controlled access ECRF for the duration of the project. Paper copies will be shredded. Should a full RCT be developed from this project participant data and samples will be transferred and used for analysis in the larger study. If at the end of this study the RCT has not yet been commenced, remaining samples and data will be transferred for safe keeping to the Peninsula Research Bank (PRB).

Sample analysis: Blood samples will be analysed for HbA1c, C-peptide and islet autoantibodies (GAD, IA2 and ZnT8) on site at the RD&E NHS FT blood sciences department. DNA will be extracted and stored for genetic testing if appropriate.

Primary Outcome measures:Time to optimum treatment following diagnosis. Optimum treatment will be determined at 3 year follow up on the basis of whether insulin is required or not (using C peptide testing if on insulin and HbA1c testing if not on insulin). If insulin is not required then the optimum treatment will be determined using the treatment guidelines for T2D or the subtype of MODY diagnosed. Treatment will be recorded 6-monthly up to 3 years.

Secondary outcome measures: Mean glycaemic control over the first 3y after diagnosis, patient satisfaction, number of hypos, weight change.

Statistics and Power Calculations The aim of this study is to determine feasibility for a future RCT, not to determine clinical differences. The investigators have therefore taken a pragmatic approach based on the number of potential recruits available over a one year period. The investigators estimate 220 people are diagnosed per year in Exeter and surrounding area. The investigators will invite all patients who fulfil the entry criteria to participate. This will enable us to determine a realistic recruitment rate and obtain estimates of rates of misclassification to inform the full RCT. Therefore, analysis will be restricted to descriptive statistics only

Ethical considerations: The investigators have discussed the potential ethical considerations with members of our PRB steering committee and addressed them as follows:

Blood sampling: a routine part diabetes care, may result in slight pain and bruising, risks minimized by sampling undertaken by staff experienced in venepuncture procedures. Patient burden: participation involves 2 blood samples (3 years apart) and 5 follow up contacts over the 3 year period (via participant choice of phone/e-mail/text). This was not considered unduly burdensome. Immediate/delayed ODS feedback: following considerable discussion around the acceptability of immediate or delayed feedback of results from the ODS, our lay members felt that considering all participants would receive treatment based on current clinical and NICE guidelines the delay in feedback of ODS results would be acceptable.

Subject Withdrawal: Subjects will be informed that they are free to withdraw from the study at any time up until the samples and data are coded but not anonymised. When samples are fully anonymised, the participants will still be able to withdraw but their samples and associated data will be retained for use in analysis.

Study Management:The study will be managed by the National Institute of Health s Research (NIHR) Exeter Clinical Research Facility providing infrastructure support and facilitate recruitment and sample collection.

Timescale: 4 years. This is a relatively long time for a pilot study and is necessary to enable data collection from each participant, over a 3 year period, to provide a clinically relevant definition of optimal treatment.

All costs will be met by existing research funding:

Sample analysis costs (HbA1c/Serum c-peptide, islet autoantibodies (GAD, IA2 and ZnT8) and Genotyping where appropriate) will be covered by the CI's existing Welcome Trust senior Investigator award. Service support costs will be provided by the NIHR Exeter Clinical Research Facility.

Project development and user involvement: The study team will have access to the user representative group of the NIHR Exeter Clinical Research Facility (ECRF). In keeping with the NHS Patient Carer and Public Involvement (PCPI) strategy the ECRF invites user representatives to contribute to the development of various projects within its portfolio. These individuals have agreed to maintain contact and regular meetings have been established at which researchers discuss the development of current projects within the ECRF.

Reporting adverse effects: This is a low risk study and it is not anticipated that participants involved in this project will be subject to adverse effects, other than slight bruising from blood sample collection. The CI will be informed of any adverse effects within 24 hours and they will be reported following local NHS R&D SOPs with a copy of any adverse event form stored in the project site file.

Participant Feedback: Depending on the randomization arm feedback from the ODS will be fed back to participants and their GP immediately or at the end of the study. Should any biochemistry immunological or genetic result potentially impact on clinical care, the results will be initially discussed with the ECRF Clinical Director and a decision may be made to contact that individual participants GP or healthcare team. A statement to this effect is included in the consent form.

Dissemination/implementation of research: Results will be written up and submitted for publication in a peer-reviewed journal. Abstracts will be submitted to national and international conferences.

Potential impact and benefit of the research: short term- the investigators hope to obtain the necessary information to conduct a definitive RCT. Longer term-evidence that the ODS can improve diagnosis and treatment for patients diagnosed with diabetes will lead to improved treatment and quality of life for patients and a reduction in the NHS costs associated with inappropriate treatment and monitoring and complication rates.

End of Study: the study will finish when all initial and follow up data has been collected and analysed on all participants.

ELIGIBILITY:
Inclusion Criteria:

* Recent clinical diagnosis of Diabetes (the working definition of recent will initially be within 3 months, but this may be modified if required).
* Aged 18 - 50 yrs of age at diagnosis.
* Able and willing to provide informed consent

Exclusion Criteria:

* Gestational diabetes
* Known secondary diabetes
* Unable/unwilling to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08-28 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Time to optimum treatment following diagnosis. | 3 years
  Optimum treatment will be determined at 3 year follow up on the basis of whether insulin is required or not (using C peptide testing if on insulin and HbA1c testing if not on insulin). If insulin is not required then the optimum treatment will be determined using the treatment guidelines for T2D or the subtype of MODY diagnosed. Treatment will be recorded 6-monthly up to 3 years.

SECONDARY OUTCOMES:
Mean glycaemic control | 3 years
  Mean glycaemic control over the first 3y after diagnosis, patient satisfaction, number of hypos, weight change.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Hattersley, Professor, Study Director — RD&E NHS FT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shields BM, Hicks S, Shepherd MH, Colclough K, Hattersley AT, Ellard S. Maturity-onset diabetes of the young (MODY): how many cases are we missing? Diabetologia. 2010 Dec;53(12):2504-8. doi: 10.1007/s00125-010-1799-4. Epub 2010 May 25. PMID 20499044
- [Result] Stone MA, Camosso-Stefinovic J, Wilkinson J, de Lusignan S, Hattersley AT, Khunti K. Incorrect and incomplete coding and classification of diabetes: a systematic review. Diabet Med. 2010 May;27(5):491-7. doi: 10.1111/j.1464-5491.2009.02920.x. PMID 20536944
- [Result] Seidu S, Davies MJ, Mostafa S, de Lusignan S, Khunti K. Prevalence and characteristics in coding, classification and diagnosis of diabetes in primary care. Postgrad Med J. 2014 Jan;90(1059):13-7. doi: 10.1136/postgradmedj-2013-132068. Epub 2013 Nov 13. PMID 24225940
- [Result] McDonald TJ, Colclough K, Brown R, Shields B, Shepherd M, Bingley P, Williams A, Hattersley AT, Ellard S. Islet autoantibodies can discriminate maturity-onset diabetes of the young (MODY) from Type 1 diabetes. Diabet Med. 2011 Sep;28(9):1028-33. doi: 10.1111/j.1464-5491.2011.03287.x. PMID 21395678
- [Result] Shields BM, McDonald TJ, Ellard S, Campbell MJ, Hyde C, Hattersley AT. The development and validation of a clinical prediction model to determine the probability of MODY in patients with young-onset diabetes. Diabetologia. 2012 May;55(5):1265-72. doi: 10.1007/s00125-011-2418-8. Epub 2012 Jan 5. PMID 22218698